CLINICAL TRIAL: NCT06397196
Title: Effects of Laser Guided Cervical Proprioceptive Exercises on Pain, Range of Motion, Cervical Position Sense and Functional Disability in Patients With Cervical Radiculopathy
Brief Title: Effects of Laser Guided Cervical Proprioceptive Exercises in Patients With Cervical Radiculopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/02105
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Range of motion; Joint Sense Position; Neck Pain; Cervical Proprioception; Neck Disability
MeSH Terms: conditions — Radiculopathy; Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Guided Proprioceptive Exercises + Routine therapy (Experimental): Participants in Group A will receive Laser guided Proprioceptive exercises with routine physical therapy on alternate days (3 days a week) for 3 weeks. total number of sessions will be 9
  Interventions: Other: Laser guided proprioceptive exercises; Other: Routine Physical therapy
- Routine Therapy (Active Comparator): Participants in Group B will receive routine physical therapy on alternate days (3 days a week) for 3 weeks. Total number of sessions will be 9.
  Interventions: Other: Routine Physical therapy

INTERVENTIONS:
Other: Laser guided proprioceptive exercises — Participants will receive Laser guided Proprioceptive exercises on alternate days (3 days a week) for 3 weeks. Total number of sessions will be 9
  Arms: Laser Guided Proprioceptive Exercises + Routine therapy
Other: Routine Physical therapy — Participants will receive routine physical therapy on alternate days (3 days a week) for 3 weeks. Total number of sessions will be 9

SUMMARY:
Cervical radiculopathy is a peripheral nervous system condition characterized by pathology of the cervical nerve root. Laser guided proprioceptive exercises shows positive impact in improving Joint sense error. The aim of this study is to investigate how proprioceptive exercises laser guided exercises, in addition to conventional exercises, affect cervical range of motion, pain, functional disability, and joint position sense error in patients with cervical radiculopathy. This randomized Controlled trial will be conducted at Islam central hospital, Sialkot. The sample size will consist of 52 participants. Participants who meet the inclusion criteria will be taken through a non-probability convenience sampling technique. 26 participants will be assigned to the group A and 26 participants to group B. Group A will receive laser guided exercises along with routine physical therapy whereas Group B will only receive routine physical therapy. All participants will receive a 50-minute session daily, 3 times a week for 3 weeks. Data will be collected using various assessment tools, Numeric pain rating scale will be use to assess the Pain, Bubble in-clinometer to assess Cervical range of motion, Laser tracker to assess Joint sense position error and Neck disability Index to assess functional disability. Pre-intervention assessment will be conducted before starting the treatment protocol and post assessment after 4 weeks of treatment.

DETAILED DESCRIPTION:
Cervical radiculopathy is a peripheral nervous system condition characterized by pathology of the cervical nerve root. Patients with cervical radiculopathy frequently appear with severe neck and arm pain as well as impaired functionality. Laser guided proprioceptive exercises shows positive impact in improving Joint sense error. The aim of this study is to investigate how proprioceptive exercises laser guided exercises, in addition to conventional exercises, affect cervical range of motion, pain, functional disability, and joint position sense error in patients with cervical radiculopathy.

This randomized Controlled trial will be conducted at Islam Central Hospital, Sialkot. The sample size will consist of 52 participants. Participants who meet the inclusion criteria will be taken through a non-probability convenience sampling technique. Participants will be randomly allocated to two groups using lottery methods. 26 participants will be assigned to the group A and 26 participants to group B. Group A will receive laser guided exercises along with routine physical therapy whereas Group B will only receive routine physical therapy. All participants will receive a 50-minute session daily, 3 times a week for 3 weeks.

Data will be collected using various assessment tools, Numeric pain rating scale will be use to assess the Pain, Bubble in-clinometer to assess Cervical range of motion, Laser tracker to assess Joint sense position error and Neck disability Index to assess functional disability. Pre-intervention assessment will be conducted before starting the treatment protocol and post assessment after 4 weeks of treatment. Data analysis will be performed using IBM SPSS version 26. Statistical significance will be set at P ≤ 0.05.The normality of data will be assessed through the Shapiro-Wilk test. The independent t-test will be used for between-group analysis, while for within-group analysis, paired T-test will be used. The difference between pre-treatment and post-treatment readings will be calculated by paired sample t-test for parametric data, whereas for non-parametric data, the Wilcoxon test will be used.

Keywords: Cervical Radiculopathy, Cervical Proprioception, Cervical joint position sense, Cervical Range of motion, Joint sense error, Neck disability index

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 55 years.
* Both Genders.
* Patients with positive Spurling test .
* Patients with positive Distraction test .
* Radicular Symptoms in Upper Extremity. (Pain, tingling or numbness in fingers and hand, weakness in arms, shoulders and hand)
* Numeric pain rate scale 3 to 7 (moderate)

Exclusion Criteria:

* Patients with cervical surgery.
* Congenital anomalies involving the cervical spine.
* Any neurological disease (e.g, cerebellar disorders, multiple sclerosis, Parkinson's disease, syringomyelia)
* Specific cause of cervical pain with previous medical diagnosis (e.g., traumatic, rheumatic or systemic pathology)
* Known or suspected vestibular pathology, dizziness, sensory nerve pathways or vascular disorders (e.g., migraine, hypertension)
* Patients suffering from Vertigo , and Vertebro basilar insufficiency (VBI).

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale. | 3 weeks
  A numerical pain rating scale (NPRS) will be used to gauge the severity of neck pain. This is an 11-point scale, where 0 is the least amount of pain (for example, "no pain") and 10 is the greatest amount of pain.
Bubble In-clinometer | 3 weeks
  Cervical Range of motion will be measured using a Bubble In-clinometer. The CROM measurements were taken while flexion, extension, left and right side bending, and left and right rotation.
Neck Disability index | 3 weeks
  We will measure the neck disability associated with pain using the neck disability index. (NDI-PT), which is valid and reliable with excellent internal consistency.
  it consists of 10 items scored out of 5. Maximum total Score = 50 A score of 0-4 is interpreted as no neck disability, 5-14 as mild, 15-24 as moderate, 25-34 as severe, and over 34 as complete neck disability.
Cervical Joint position sense error | 3 weeks
  To measure the joint position sense error.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.phill, Principal Investigator — Riphah Intenational University
Locations (1):
- Islam Central Hospital., Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L, Knezevic NN, Navani A, Christo PJ, Limerick G, Calodney AK, Grider J, Harned ME, Cintron L, Gharibo CG, Shah S, Nampiaparampil DE, Candido KD, Soin A, Kaye AD, Kosanovic R, Magee TR, Beall DP, Atluri S, Gupta M, Helm Ii S, Wargo BW, Diwan S, Aydin SM, Boswell MV, Haney BW, Albers SL, Latchaw R, Abd-Elsayed A, Conn A, Hansen H, Simopoulos TT, Swicegood JR, Bryce DA, Singh V, Abdi S, Bakshi S, Buenaventura RM, Cabaret JA, Jameson J, Jha S, Kaye AM, Pasupuleti R, Rajput K, Sanapati MR, Sehgal N, Trescot AM, Racz GB, Gupta S, Sharma ML, Grami V, Parr AT, Knezevic E, Datta S, Patel KG, Tracy DH, Cordner HJ, Snook LT, Benyamin RM, Hirsch JA. Epidural Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Comprehensive Evidence-Based Guidelines. Pain Physician. 2021 Jan;24(S1):S27-S208. PMID 33492918
- [Background] Borrella-Andres S, Marques-Garcia I, Lucha-Lopez MO, Fanlo-Mazas P, Hernandez-Secorun M, Perez-Bellmunt A, Tricas-Moreno JM, Hidalgo-Garcia C. Manual Therapy as a Management of Cervical Radiculopathy: A Systematic Review. Biomed Res Int. 2021 Jun 3;2021:9936981. doi: 10.1155/2021/9936981. eCollection 2021. PMID 34189141
- [Background] Savva C, Korakakis V, Efstathiou M, Karagiannis C. Cervical traction combined with neural mobilization for patients with cervical radiculopathy: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:279-289. doi: 10.1016/j.jbmt.2020.08.019. Epub 2020 Sep 2. PMID 33992259
- [Background] Maharaj RG, Motilal S, Khan R, Rampersad F. A No-Cost, Bedside, Self-Traction Maneuver for Relief From Chronic Cervical Radiculopathy: A Case Report. Cureus. 2023 Aug 23;15(8):e43963. doi: 10.7759/cureus.43963. eCollection 2023 Aug. PMID 37746470
- [Background] Mendes-Fernandes T, Puente-Gonzalez AS, Marquez-Vera MA, Vila-Cha C, Mendez-Sanchez R. Effects of Global Postural Reeducation versus Specific Therapeutic Neck Exercises on Pain, Disability, Postural Control, and Neuromuscular Efficiency in Women with Chronic Nonspecific Neck Pain: Study Protocol for a Randomized, Parallel, Clinical Trial. Int J Environ Res Public Health. 2021 Oct 12;18(20):10704. doi: 10.3390/ijerph182010704. PMID 34682453
- [Background] Pennetti A. A multimodal physical therapy approach utilizing the Maitland concept in the management of a patient with cervical and lumbar radiculitis and Ehlers-Danlos syndrome-hypermobility type: A case report. Physiother Theory Pract. 2018 Jul;34(7):559-568. doi: 10.1080/09593985.2017.1422207. Epub 2018 Jan 8. PMID 29308941